CLINICAL TRIAL: NCT04302376
Title: Thrombotic Complications After Central Venous Catheterization: a Prospective Observational Study
Brief Title: Thrombotic Complications After Central Venous Catheterization
Acronym: TARZAN
Status: Completed | Type: Observational
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Jasper M Smit, MD, Prinicpal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: 2019.575
Record Dates: First submitted 2019-11-25; First posted 2020-03-10 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Central Venous Catheter Thrombosis
Keywords: central venous catheter; catheter-related thrombosis; CVC; ultrasound
MeSH Terms: conditions — Upper Extremity Deep Vein Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Catheter-related thrombosis: The presence of occlusive or nonocclusive thrombus in the insertion vein ad identified on Doppler and compression ultrasonography and compression ultrasound.
  Interventions: Diagnostic Test: Cather-related thrombosis ultrasonography
- No catheter-related thrombosis: The absence of occlusive or nonocclusive thrombus in the insertion vein ad identified on Doppler and compression ultrasonography and compression ultrasound.
  Interventions: Diagnostic Test: Cather-related thrombosis ultrasonography

INTERVENTIONS:
Diagnostic Test: Cather-related thrombosis ultrasonography — Doppler and compression ultrasound to detect catheter-related thrombosis

SUMMARY:
Rationale: Complications related to central venous catheterization are mechanical, infectious or thrombotic in origin. Potential complications of catheter-related thrombosis are not insubstantial and include pulmonary embolism, post-thrombotic syndrome or thrombophlebitis. Prevalence and incidence of catheter-related thrombosis at the intensive care unit is unclear and treatment, especially of asymptomatic thrombosis, remains ambiguous. Therefore a study is warranted that evaluates the prevalence and incidence of catheter-related thrombosis and investigates its potential consequences. We hypothesize that the incidence of catheter-related thrombosis is 5-15%.

Objective: To assess the prevalence and incidence of symptomatic and asymptomatic catheter-related thrombosis.

DETAILED DESCRIPTION:
INTRODUCTION AND RATIONALE

Since its introduction, central venous catheter (CVC) use has been increasing and is now indispensable in modern-day medical practice. Besides its imperative use in critically ill patients, there are multiple complications associated with central venous catheterization. Complications are mechanical, infectious or thrombotic in origin. There is a growing body of literature that recognises the potential deleterious consequences of catheter-related bloodstream infections and this complication has been the main focus of research. In contrast, despite catheter-related thrombosis being a well-known complication and accounting for approximately 15 percent of all venous thromboses in ICU patients, its exact incidence and potential consequences in ICU patients remain unclear.

Histologically, due to intravascular movement of the CVC focal areas of endothelial injury in the vein wall adjacent to the catheter occur. Simultaneously, a fibrin sheath grows along the catheter surface from the venotomy site. The fibrin sheath, in combination with endothelial injury and a decreased blood flow around the catheter triggers the development of catheter-related thrombosis. The formed thrombus can gradually increase in size until there is occlusion of the vein and, subsequently, symptoms of localized swelling, pain, tenderness and erythema along the course of the vein may occur.

Up to now CVCs are removed without routinely investigating the presence of catheter-related thrombosis. Therefore, its exact incidence is ambiguous and among asymptomatic patients the natural course of catheter-related thrombosis remains uncertain. Potential consequences of catheter-related thrombosis are not insubstantial; they include pulmonary embolism, post-thrombotic syndrome, thrombophlebitis, treatment delay, and loss of venous access. However, a study by Jones et al., conducted in children who received a CVC in the internal jugular or femoral vein, showed low risk for developing short and long-term sequalae after catheter-related thrombosis. Moreover, another study by White et al. showed no increased risk of developing pulmonary embolism after central venous catheter placement.

To date, there is no consensus regarding treatment of catheter-related thrombosis in ICU patients. In case it becomes symptomatic, guidelines for lower extremity deep vein thrombosis are followed and patients are treated accordingly. However, in case catheter-related thrombosis is an accidental find and remains asymptomatic, treatment is more controversial. Some physicians decide to treat it with anticoagulants, whereas others do not treat it at all.

If we take into account that the natural history of catheter-related thrombosis remains unclear in adult ICU patients and its treatment is even more controversial, a study is warranted that investigates the incidence and potential sequelae of catheter-related thrombosis. The primary aim of this study is to evaluate the incidence of catheter-related thrombosis in adult ICU patients and to investigate its relationship with potentially hazardous sequelae.

OBJECTIVES

Primary Objective:

- To evaluate the prevalence and incidence of catheter-related thrombosis in adult ICU patients

Secondary Objectives:

* To investigate the correlation between catheter-related thrombosis and catheter-related infections
* To identify potential risk factors associated with catheter-related thrombosis
* To investigate the association of catheter-related thrombosis with potential sequalae

ELIGIBILITY:
Inclusion Criteria:

* Central venous cannulation of the internal jugular vein, subclavian vein, or femoral vein
* ≥ 48 hours catheter indwelling time

Exclusion Criteria:

* Removal of the CVC within 48 hours after placement
* Pre-existent thrombosis at vein of insertion site
* Discharge of patients from ICU with CVC in situ
* Inability to perform compression and colour Doppler ultrasound evaluation of cannulated vein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (≥18 years) patients admitted to the ICU receiving a CVC at the ICU, are admitted to the ICU after surgery and received a CVC in advance, or are admitted from the emergency department and have a CVC placed just before ICU admission.
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence and prevalence of catheter-related thrombosis | Date of central venous catheter insertion until date of catheter removal, assessed up to 28 days after CVC insertion
  Prevalence and incidence of catheter-related thrombosis per 1000 catheter days. Catheter-related thrombosis will be divided into asymptomatic and symptomatic catheter-related thrombosis:
  Asymptomatic thrombosis: the presence of occlusive or nonocclusive thrombus in insertion vein as identified on Doppler and compression ultrasonography and the absence of any clinical signs or symptoms of thrombosis of the area Symptomatic thrombosis: The presence of occlusive or nonocclusive thrombus in the insertion vein as identified on Doppler and compression ultrasonography and the presence of at least 1 of the following signs or symptoms: swelling, pain, redness, or discoloration of the area; dysfunction of the CVC.

SECONDARY OUTCOMES:
Correlation of catheter-related thrombosis with catheter-related infections | Date of central venous catheter insertion until date of catheter removal, assessed up to 28 days after CVC insertion
  Catheter-related infections will be divided into three subgroups:
  Local catheter infection: clinical signs of infection at CVC insertion site (redness, pus) in combination with a positive culture from the skin and/or pus at the insertion site Clinical suspicion of catheter infection: one or more of the following: local infection; fever of unknown origin, with CVC present for ≥ 3 days; positive blood cultures without clear focus of infection at other site; normalization of temperature after CVC removal Catheter-related bloodstream infection (CRBSI): Clinical suspicion of infection (fever, chills, unexplained leukocytosis, hypotension, tachycardia etc.) with no clear focus apart from the central line, or signs of local infection around the insertion site, in combination with a positive culture from a catheter segment and at least one positive blood culture of the same pathogen. The blood sample must be drawn from a different location than from the potentially infected central line.
Risk factors associated with catheter-related thrombosis. | Date of central venous catheter insertion until date of catheter removal, assessed up to 28 days after CVC insertion
  Potential risk factors are identified using previously published literature or are theoretically based on Virchow's triad: patient characteristics, CVC-tip location, lumen diameter, number of lumens, insertion site, duration of insertion procedure, arterial puncture, vein diameter, (lumen diameter/vein diameter) indwelling time, number of cannulation attempts, elective or emergency insertion and experience of investigator inserting the CVC.
Association of catheter-related thrombosis with development of pulmonary embolism | Date of central venous catheter removal up to 1 month of follow up, hospital discharge or death
  Pulmonary embolism as seen on CT
Association of catheter-related thrombosis with development of symptomatic thrombosis | Date of central venous catheter removal up to 1 month of follow up, hospital discharge or death
  Symptomatic thrombosis: the presence of occlusive or nonocclusive thrombus in the insertion vein as identified on Doppler and compression ultrasonography and the presence of at least 1 of the following signs or symptoms: swelling, pain, redness, or discoloration of the area; dysfunction of the CVC.
Association of catheter-related thrombosis with development of suppurative (septic) thrombophlebitis. | Date of central venous catheter removal up to 1 month of follow up, hospital discharge or death
  Suppurative thrombophlebitis: persistent bacteraemia for 72 hours after catheter removal despite appropriate antimicrobial therapy in combination with symptomatic or asymptomatic thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Coded data can be shared with other researchers after publication of study

REFERENCES:
- [Background] Parienti JJ, Mongardon N, Megarbane B, Mira JP, Kalfon P, Gros A, Marque S, Thuong M, Pottier V, Ramakers M, Savary B, Seguin A, Valette X, Terzi N, Sauneuf B, Cattoir V, Mermel LA, du Cheyron D; 3SITES Study Group. Intravascular Complications of Central Venous Catheterization by Insertion Site. N Engl J Med. 2015 Sep 24;373(13):1220-9. doi: 10.1056/NEJMoa1500964. PMID 26398070
- [Background] Jones S, Butt W, Monagle P, Cain T, Newall F. The natural history of asymptomatic central venous catheter-related thrombosis in critically ill children. Blood. 2019 Feb 21;133(8):857-866. doi: 10.1182/blood-2018-05-849737. Epub 2018 Oct 30. PMID 30377196
- [Background] Wall C, Moore J, Thachil J. Catheter-related thrombosis: A practical approach. J Intensive Care Soc. 2016 May;17(2):160-167. doi: 10.1177/1751143715618683. Epub 2015 Dec 3. PMID 28979481